CLINICAL TRIAL: NCT00440531
Title: A Study in Healthy Adults of the Safety, Tolerability, and Immunogenicity of Recombinant Hepatitis B Vaccine Manufactured With a Modified Process
Brief Title: Study of Recombinant Modified Process Hepatitis B Vaccine in Older Adults (V232-059)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V232-059; 2007_516
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2009-03-31 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): RECOMBIVAX HB™
  Interventions: Biological: Comparator: RECOMBIVAX HB™ Hepatitis B Vaccine (Recombinant)
- 2 (Experimental): Modified Process Hepatitis B Vaccine
  Interventions: Biological: Comparator: Modified Process Hepatitis B Vaccine (Experimental)
- 3 (Active Comparator): ENGERIX-B™
  Interventions: Biological: Comparator: ENGERIX-B™ (currently licensed product)

INTERVENTIONS:
Biological: Comparator: RECOMBIVAX HB™ Hepatitis B Vaccine (Recombinant) — RECOMBIVAX HB™ (currently licensed product) given IM (Intramuscular) in 3 doses of 10 mcg (micrograms)/1.0 mL each over 6 months.
  Arms: 1
Biological: Comparator: Modified Process Hepatitis B Vaccine (Experimental) — Modified Process Hepatitis B Vaccine (Experimental) given IM (Intramuscular) in 3 doses of 10 mcg (micrograms)/1.0 mL each over 6 months.
  Arms: 2
Biological: Comparator: ENGERIX-B™ (currently licensed product) — ENGERIX-B™ given IM (Intramuscular) in 3 doses of 20 mcg (micrograms)/1.0 mL each over 6 months.
  Arms: 3

SUMMARY:
The purpose of this trial is to determine if there is an improvement in the immune response of older adults over 50 years of age using a modified process hepatitis B vaccine and a currently licensed hepatitis B vaccine (RECOMBIVAX HB™).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female older adults greater than or equal to 50 years of age

Exclusion Criteria:

* Any adult with a history of previous hepatitis B infection
* A history of vaccination with any hepatitis B vaccine
* Recent (<72 hours) history of febrile illness (oral temperature =37.8ºC/=100.0ºF)
* Known or suspected hypersensitivity to any component of RECOMBIVAX HB™ or ENGERIX-B™ (e.g., aluminum, yeast)
* Recent administration (within 3 months prior to first injection with the study vaccine) of hepatitis B immune globulin (HBIG), serum immune globulin, or any other blood-derived product
* Receipt of licensed inactivated vaccines within 14 days prior to first injection with the study vaccine
* Receipt of licensed live virus vaccines within the 30 days prior to injection with the study vaccine
* Receipt of investigational drugs or other investigational vaccines within 3 months prior to first injection with the study vaccine
* Known or suspected impairment of immunologic function or recent use of immunomodulatory medications (e.g., systemic corticosteroids). Does not include topical and inhaled steroids
* Pregnant women, nursing mothers, and women planning to become pregnant within the study period
* Any condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Gilbert CL, Klopfer SO, Martin JC, Schodel FP, Bhuyan PK. Safety and immunogenicity of a modified process hepatitis B vaccine in healthy adults >/=50 years. Hum Vaccin. 2011 Dec;7(12):1336-42. doi: 10.4161/hv.7.12.18333. Epub 2011 Dec 1. PMID 22185811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27-Nov-2006 (First Participant Enrolled in Study) to 26-Nov-2007 (Last Participant had their Last Visit). This study was conducted at 22 sites: 10 in Canada, 2 in Denmark, 5 in Sweden, and 5 in the United Kingdom.
Pre-assignment Details: In the Modified Process group, 2 participants were randomized but not vaccinated: 1 participant withdrew consent, and 1 participant had an SAE (Serious Adverse Experience) of hypertension prior to vaccination.
Groups:
- Modified Process Hepatitis B Vaccine: Modified Process Hepatitis B Vaccine, 10 µg (micrograms)
- RECOMBIVAX-HB™: RECOMBIVAX-HB™, 10 µg (micrograms)
- ENGERIX-B™: ENGERIX-B™, 20 µg (micrograms)
Period: Overall Study
Arm/Group | Modified Process Hepatitis B Vaccine | RECOMBIVAX-HB™ | ENGERIX-B™
Started | 185 | 183 | 172
Vaccination 1 | 183 | 183 | 172
Vaccination 2 | 181 | 182 | 171
Vaccination 3 | 176 | 178 | 166
Completed | 175 | 178 | 165
Not Completed | 10 | 5 | 7
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Lost to Follow-up | 4 | 3 | 5
Not completed — see pre-assignment details | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Process Hepatitis B Vaccine | RECOMBIVAX-HB™ | ENGERIX-B™ | Total
Number analyzed (Participants) | 183 | 183 | 172 | 538
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (7.9) | 60.4 (7.6) | 59.8 (6.5) | 60.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 73 | 260
  Male | 90 | 89 | 99 | 278

OUTCOME MEASURES:

1. Primary Outcome: The Number of Seroresponders to the Modified Process Hepatitis B Vaccine and RECOMBIVAX HB™ (Currently Licensed Vaccine)
Description: The number of participants as measured by the seroprotection rate (anti-hepatitis B surface antibodies greater than or equal to 10 mIU/mL). Anti-HBs (Antibodies against hepatitis B surface antigen) titers were measured from blood samples taken at Day 1 (prior to the first vaccination) and at Month 7 (1 month after the third vaccination).
Time Frame: 7 months (1 month after third vaccination)
Population: Per-protocol Population. The Per-protocol Population is defined as the participants that were able to complete the study as defined by the protocol.
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | RECOMBIVAX-HB™
Number analyzed (Participants) | 152 | 147
Participants | 115 | 100
Statistical Analysis 1: Comparison: Modified Process Hepatitis B Vaccine; No hypothesis is being tested. The purpose of the primary analysis is to estimate the seroprotection rate (percentage of subjects with anti-HBs >=10mIU/mL) in each group at 1 month post vaccination 3, among subjects who were seronegative at baseline; Test type: Superiority or Other; single-group percentage = 75.70, 95% CI [68 to 82.20]
Statistical Analysis 2: Comparison: RECOMBIVAX-HB™; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; single-group percentage = 68, 95% CI [59.80 to 75.50]

2. Secondary Outcome: The Number of Seroresponders to ENGERIX-B™ (Currently Licensed Vaccine)
Description: as for outcome 1
Time Frame: 7 months (1 month after third vaccination)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ENGERIX-B™
Number analyzed (Participants) | 144
Participants | 121
Statistical Analysis 1: Comparison: ENGERIX-B™; No hypothesis is being tested. The purpose of the secondary analysis is to estimate the seroprotection rate (percentage of subjects with anti-HBs >=10mIU/mL) for ENGERIX-B™ at 1 month post vaccination 3, among subjects who were seronegative at baseline; Test type: Superiority or Other; Single-Group Percentage = 84, 95% CI [77 to 89.60]

3. Secondary Outcome: The Total Number of Participants With One or More Injection-site Adverse Experiences
Time Frame: Days 1-5 After Any Vaccination
Population: Safety Analysis Set - defined as all participants who received at least one injection of vaccine and who had a safety follow-up.
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | RECOMBIVAX-HB™ | ENGERIX-B™
Number analyzed (Participants) | 182 | 183 | 171
Participants | 103 | 115 | 107

4. Secondary Outcome: The Total Number of Participants With a Maximum Temperature >=100.0F/37.8C
Time Frame: Day 1-5 After Vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | RECOMBIVAX-HB™ | ENGERIX-B™
Number analyzed (Participants) | 182 | 183 | 171
Participants | 2 | 3 | 3

5. Secondary Outcome: The Total Number of Participants With Serious Vaccine-Related Clinical Adverse Experiences
Time Frame: During Entire Study Period (from first vaccination until the participant completes or discontinues: up to 7 months)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Modified Process Hepatitis B Vaccine | RECOMBIVAX-HB™ | ENGERIX-B™
Number analyzed (Participants) | 182 | 183 | 171
Participants | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.